CLINICAL TRIAL: NCT03955757
Title: Using Boot Camp Translation to Address Rural Disparities in Adolescent Vaccination
Acronym: RADVax
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Colorado, Denver (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 18-1588; U01IP001091 (NIH)
Record Dates: First submitted 2019-05-13; First posted 2019-05-20 (Actual); Last update posted 2022-08-16 (Actual); Status verified 2022-08

CONDITIONS: Primary Prevention
Keywords: Immunization; Boot Camp Translation; Adolescent

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The study team data analyst will be provided with blinded data.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Boot Camp Translation (Experimental): Intervention communities will undergo the Boot Camp Translation process.
  Interventions: Behavioral: Boot Camp Translation
- Control (Active Comparator): Control communities will behave as usual
  Interventions: Other: Control

INTERVENTIONS:
Behavioral: Boot Camp Translation — Communities in the intervention arm will participate in the Boot Camp translation process, where stakeholders will come together to develop and implement locally relevant materials to promote adolescent vaccination.
  Arms: Boot Camp Translation
Other: Control — No intervention. Communities will continue to behave as usual.
  Arms: Control

SUMMARY:
The overall goal of this project is to implement the Boot Camp Translation process to develop a replicable approach for increasing adolescent vaccine uptake that can be adaptable and feasible to use in rural settings more broadly.

DETAILED DESCRIPTION:
Boot Camp Translation (BCT) is a process to identify strategies that help communities improve health. It is a 6-month, facilitated, iterative community engagement process that brings together relevant stakeholders to develop and implement locally meaningful messages, materials, and strategies for health topics of interest.

This is a novel community engagement process that has a proven ability to result in meaningful and impactful strategies to improve compliance with recommended health behaviors in rural communities. The investigators will expand this work by testing BCT on its ability to improve vaccination with all recommend adolescent vaccines (Tdap, MenACWY, HPV, Flu).

The investigators will conduct a randomized, controlled trial in which 4 rural communities in Western Colorado will undergo BCT to develop and implement strategies to increase adolescent vaccination. Vaccination rates will be compared to 4 control communities that do not undergo BCT.

ELIGIBILITY:
Inclusion Criteria:

* Must live in one of the designated Colorado communities

Exclusion Criteria:

* Does not live in one of the designated Colorado communities

Ages: 11 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 6000 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2022-08-31 (Estimated); Study Completion 2022-08-31 (Estimated)

PRIMARY OUTCOMES:
Initiation of HPV vaccination series, 11-12 year olds | Up to 24 months
  Percent of 11-12 year olds who have received >=1 dose of the HPV vaccine by May 31,2021

SECONDARY OUTCOMES:
Completion of HPV vaccination series, 11-12 year olds | Up to 24 months
  Percent of 11-12 year olds with >=2 doses of the HPV vaccine by May 31,2021
Initiation of HPV vaccination series, 13-17 year olds | Up to 24 months
  Percent of 13-17 year olds who have received >=1 dose of the HPV vaccine by May 31,2021
Completion of HPV vaccination series, 13-17 year olds | Up to 24 months
  Percent of 13-17 year olds who have completed the HPV vaccine series (2 or 3 doses, depending on age of initiation) by May 31,2021
Receipt of Tdap vaccine, 11-12 year olds | Up to 24 months
  Percent of 11-12 year olds who have received Tdap vaccine by May 31,2021
Receipt of Tdap vaccine, 13-17 year olds | Up to 24 months
  Percent of 13-17 year olds who have received Tdap vaccine by May 31,2021
Receipt of MCV vaccine, 11-12 year olds | Up to 24 months
  Percent of 11-12 year olds who have received >=1 dose of MCV vaccine by May 31,2021
Receipt of MCV vaccine, 13-17 year olds | Up to 24 months
  Percent of 13-17 year olds who have received >=1 dose of MCV vaccine by May 31,2021

OTHER OUTCOMES:
Receipt of influenza vaccine | Up to 24 months
  Percent of 11-17 year olds who receive the influenza vaccine between Sept 2020 and May 2021

CONTACTS AND LOCATIONS:
Overall Officials: Sean T O'Leary, MD, Principal Investigator — University of Colorado, Denver; Amanda Dempsey, MD, PhD, MPH, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Anschutz Medical Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cataldi JR, Suresh K, Brewer SE, Perreira C, Nederveld A, Skenadore A, Furniss A, Williams C, Severson R, Dempsey AF, O'Leary ST. Boot Camp Translation using Community-Engaged messaging for adolescent Vaccination: A Cluster-Randomized trial. Vaccine. 2024 Feb 15;42(5):1078-1086. doi: 10.1016/j.vaccine.2024.01.042. Epub 2024 Jan 21. PMID 38253469